CLINICAL TRIAL: NCT00868751
Title: Single Patient Use of Tocilizumab for Treatment of Steroid Dependent, Active Systemic Onset Juvenile Idiopathic Arthritis
Brief Title: Single Patient Use of Tocilizumab in Systemic Onset Juvenile Idiopathic Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Hyperintensities of unclear etiology on brain MRI. Follow up revealed no progression.
Sponsor: Tufts Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-PRHEU-TCZ-01
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Arthritis, Juvenile Rheumatoid; Still's Disease, Juvenile Onset
Keywords: Antibodies, Monoclonal; Interleukin 6
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tocilizumab (Experimental): Single arm study - treatment only
  Interventions: Biological: tocilizumab

INTERVENTIONS:
Biological: tocilizumab — Initial therapy: Tocilizumab dosed by body weight (8mg/kg based on body weight ≥ 30kg) given by intravenous infusion every two weeks for 12 weeks.
  Extension of therapy: Continuation of treatment with tocilizumab at 8mg/kg by body weight given by intravenous infusion every 2 weeks based upon achievement of Primary Objective by week 12, OR continuation of treatment with escalation of tocilizumab dose to 12mg/kg by body weight, given by intravenous infusion every two weeks, for failure to achieve ACR JIA30 at 12 weeks or ACR JIA50 response at any time after week 16.
  Other Names: Actemra, RoACTEMRA, MRA

SUMMARY:
The purpose of this study is to see if tocilizumab is safe and effective for treating systemic onset Juvenile Idiopathic Arthritis (soJIA). Another purpose is to see if tocilizumab helps reduce the amount of steroids (prednisone) needed to control symptoms of soJIA.

DETAILED DESCRIPTION:
Systemic onset Juvenile Idiopathic Arthritis (soJIA) is a type of arthritis (inflammation of the joints) that occurs with other symptoms including fever, swollen lymph nodes (glands), rash, and body aches. Because soJIA can be difficult to treat, children with soJIA can have severe problems from long-term use of steroids (prednisone). These problems include low bone density (weak bones), fractures, failure to grow properly, and large weight gain. The arthritis that occurs in soJIA often causes damage to many joints. This can make it hard to move around or do basic tasks like dressing. Also, a life-threatening illness called Macrophage Activation Syndrome (MAS) can occur when starting, stopping, or changing drugs that are used to treat soJIA.

SoJIA can be hard to treat and many children with soJIA do not respond to drugs that work for other kinds of arthritis. Research doctors have studied a chemical signal called IL-6 that the body uses to manage inflammation. This signal has been found to be very high in patients with active soJIA. A drug called tocilizumab (TCZ) has been designed to block IL-6. For about 6 years, TCZ has been tested in Japan for treating soJIA. It is now being tested in studies in the United States. These studies can have very strict rules for enrolling patients. This trial is a single-patient research study for a subject who otherwise does not meet the rules for enrollment in ongoing trials.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Juvenile Idiopathic Arthritis according to ILAR criteria (2001)
* Duration of disease ≥ 6 months since onset
* Presence of active disease as determined by the presence of at least 5 active joints, OR at least 2 active joints if receiving prednisone at a dose > 0.2 mg/kg/day or > 10 mg/day (whichever is less)
* Incomplete prior response to methotrexate treatment for at least 3 months at a minimum dose of 15 mg/M2/week, or intolerance to methotrexate
* Discontinued treatment with other biologics prior to first tocilizumab infusion, for approximately two pharmacokinetic half-lives as per specific biologic (e.g. 48 hours for anakinra, 7 days for etanercept)
* Not receiving corticosteroids, OR taking oral corticosteroids and the dose has remained stable for 1 week prior to the first tocilizumab infusion at ≤ 2 mg/kg/day prednisone or prednisolone and no more than 80 mg/day

Exclusion Criteria:

* Concomitant administration of biologic therapies
* Serum creatinine >1.5 ULN (upper limits normal)
* AST or ALT > 1.5 ULN
* Total bilirubin > 1.3 mg/dL
* Platelet count < LLN (lower limits normal)
* Hemoglobin < 6.0 g/dL
* WBC count < 5,000/mm3
* Neutrophil count < 2,000/ mm3
* Fibrinogen < LLN

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Natter, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center/Floating Hospital for Children, Boston, Massachusetts, United States

REFERENCES:
- [Background] Yokota S, Imagawa T, Mori M, Miyamae T, Aihara Y, Takei S, Iwata N, Umebayashi H, Murata T, Miyoshi M, Tomiita M, Nishimoto N, Kishimoto T. Efficacy and safety of tocilizumab in patients with systemic-onset juvenile idiopathic arthritis: a randomised, double-blind, placebo-controlled, withdrawal phase III trial. Lancet. 2008 Mar 22;371(9617):998-1006. doi: 10.1016/S0140-6736(08)60454-7. PMID 18358927
- See also: A Study of Tocilizumab in Patients With Active Systemic Juvenile Idiopathic Arthritis — http://www.clinicaltrials.gov/ct2/show/NCT00642460

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Single arm study - treatment only
  tocilizumab: Initial therapy: Tocilizumab dosed by body weight (8mg/kg based on body weight ≥ 30kg) given by intravenous infusion every two weeks for 12 weeks.
  Extension of therapy: Continuation of treatment with tocilizumab at 8mg/kg by body weight given by intravenous infusion every 2 weeks based upon achievement of Primary Objective by week 12, OR continuation of treatment with escalation of tocilizumab dose to 12mg/kg by body weight, given by intravenous infusion every two weeks, for failure to achieve ACR JIA30 at 12 weeks or ACR JIA50 response at any time after week 16.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Tocilizumab as Defined by Presence of an Equal to or Greater Than 30% Improvement in JIA Core Set (i.e. ACR JIA30 Response)
Time Frame: At week 12 of treatment versus week 0 (pretreatment)
Population: No data are available because data were not collected
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

2. Primary Outcome: Efficacy of Tocilizumab as Defined by Reduction of Oral Prednisone Dose by at Least 20%, or to Less Than 0.5mg/kg/Day, Whichever is of Lesser Daily Dose, While Maintaining an ACR JIA30 Response
Time Frame: At weeks 12 and 16 of treatment versus week 0 (pretreatment)
Population: No data are available because data were not collected
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: To evaluate the safety of tocilizumab administration in this subject
Time Frame: Ongoing, throughout 24 month study period
Population: No data are available because data were not collected
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Measurement of Laboratory Parameters of Active Disease, Specifically C-reactive Protein, Hemoglobin, Platelets, White Blood Cell Count, Ferritin, Immunoglobulins.
Description: To assess normalization of laboratory parameters of active disease, specifically C-reactive protein, hemoglobin, platelets, white blood cell
Time Frame: At weeks 8, 12, and 16 of treatment, and every 8-12 weeks thereafter
Population: No data are available because data were not collected
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Measurement of Sustained Clinical Response to Tocilizumab, Including Active Joint Count, Joints With Limited Range of Motion, and Absence of Fever or Rash.
Description: To assess sustained clinical response to tocilizumab, including active joint count, joints with limited range of motion, and absence of fever
Time Frame: At weeks 8, 12, 16 of treatment, and every 8 weeks thereafter
Population: No data are available because data were not collected
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=1)
Hyperintensities of unclear etiology on brain MRI. Follow up revealed no progression. (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes